CLINICAL TRIAL: NCT03258476
Title: Guanfacine Extended Release and Mindfulness in Traumatically Stressed Children and Adolescents Study
Brief Title: Guanfacine Extended Release and Mindfulness Skills Therapy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Contract terminated
Sponsor: UConn Health (Other)
Collaborators: Shire (Industry); Yale University (Other)
Responsible Party: Principal Investigator, Asima Zehgeer, Assistant Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-080-2
Record Dates: First submitted 2017-05-24; First posted 2017-08-23 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Stress Disorder
MeSH Terms: conditions — Stress Disorders, Traumatic | interventions — Guanfacine

STUDY DESIGN:
Intervention Model Description: The proposed study has two parts: (1) a randomized, double-blind controlled clinical trial of GXR vs. placebo for up to 7 weeks followed by, (2) 10 weeks of either GXR and Mindfulness psychotherapy (as a group or individual) or placebo and Mindfulness psychotherapy (as a group or individual).
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- GXR and Mindfulness Skills (Experimental): Guanfacine Extended Release (GXR) will be started at 1 mg/day at Week 1 and tapered up by 1 mg per week to a maximum dose of 7 mg/day by week 7 (maximum of 6 weeks on drug). GXR dosing will be flexible for the first 5 weeks of the study based upon patient response and tolerability to drug. Optimal dose will be defined as that necessary to achieve ≥ 30% reduction in symptoms and a CGI-Improvement Score ≤ 2. Upon re-evaluation at (T1) and entry into the psychotherapy protocol dosing will become fixed for the remainder of the study. Mindfulness Skills Therapy will occur for the next 10 weeks.
  Interventions: Drug: Guanfacine Extended Release; Behavioral: Mindfulness Skills Therapy
- Placebo and Mindfulness Skills (Active Comparator): Placebo will be started at "1 mg/day" at Week 1 and tapered up by "1 mg" per week to a maximum dose of "7 mg/day" by week 7 (maximum of 6 weeks on drug). Placebo dosing will be flexible for the first 5 weeks of the study based upon patient response. Optimal dose will be defined as that necessary to achieve ≥ 30% reduction in symptoms and a CGI-Improvement Score ≤ 2. Upon re-evaluation at (T1) and entry into the psychotherapy protocol dosing will become fixed for the remainder of the study. Mindfulness Skills Therapy will occur for the next 10 weeks.
  Interventions: Behavioral: Mindfulness Skills Therapy; Drug: Placebo

INTERVENTIONS:
Drug: Guanfacine Extended Release — Intuniv (guanfacine) is a prescription medicine used to treat attention deficit hyperactivity disorder (ADHD) in children who are at least 6 years old. An open-label trail of guanfacine extended release (GXR 1-4 mg/daily; Intuniv™) suggested benefits in improving behavioral and emotional regulation in children and adolescents with symptoms of traumatic stress. However, to date no controlled clinical trial has been completed assessing the effects of GXR on traumatic stress symptoms in youths
  Other Names: Intuniv
  Arms: GXR and Mindfulness Skills
Behavioral: Mindfulness Skills Therapy — Mindfulness is a therapy for anxiety and stress. Mindfulness forms of therapy involve regulation of attention, maintaining it in immediate experience, regardless of the valence and desirability of the experience. To reduce anxiety, Mindfulness encourages observing and accepting anxiety-related thoughts
Drug: Placebo — Placebo oral capsule
  Arms: Placebo and Mindfulness Skills

SUMMARY:
Teenagers are invited to take part voluntarily in a research study of a study drug known as guanfacine extended release (Intuniv™) and a type of psychotherapy called Mindfulness Skills Training which teaches people how to focus on the present moment in a nonjudgmental manner to help them cope with their stresses and worries. Teenagers are being asked to take part in this study if they have had traumatic stress related over arousal symptoms. He/she may also have difficulties with worries, anxiety, temper, aggression, quick mood changes, behavior problems, and/or difficulties with symptoms of Attention Deficit Hyperactivity Disorder (ADHD) including inattention, hyperactivity, and impulsivity with or without Posttraumatic Stress Disorder (PTSD); and is not responding adequately to his/her current treatment.

The primary purpose of the teenager's participation in this study is to help answer the following research question(s), and not to provide treatment for his or her condition:

* To investigate if Intuniv™ helps for the symptoms of traumatic stress and emotional and behavioral overarousal in children with a history of traumatic developmental stress with and without PTSD.
* To investigate if Intuniv™ helps your teenager engage with and benefit from Mindfulness Skills Training therapy
* To better understand how Intuniv™ works in the brain.
* To investigate how well your child tolerates Intuniv™ during the study.

ELIGIBILITY:
Inclusion Criteria:

* A lifetime history of traumatic stress documented by self and/or caregiver response on the youth self-report and or caregiver-report Structured Trauma-Related Experiences & Symptoms Screener (STRESS) (i.e., at least one yes response on STRESS items 1-25). AND
* A baseline STRESS total score ≥ 21 for females or a baseline STRESS total score ≥ 17 for males (STRESS items # 26-48: range of total scores: 0-69) 68 as completed by caregiver OR youth.

AND/OR

* A lifetime history of traumatic stress documented by self and/or caregiver response on the youth self-report and or caregiver-report Structured Trauma-Related Experiences & Symptoms Screener (STRESS) (i.e., at least one yes response on STRESS items 1-25). AND
* Clinically significant aggressive behavior during the preceding week assessed by a caregiver-completed Retrospective Modified Overt Aggression (R-MOAS ≥ 24).73 AND
* A baseline Clinical Global Impressions-Severity Score ≥ 4.74
* Assent of child and consent of both parents/caregivers.
* Living with a caregiver legally empowered to permit study enrollment and able to complete protocol assessments.
* English speaking
* The child is not responding to or is not tolerating well their current treatment as reported by the parent or child.
* If female and reports that she is sexually active: Is willing to take a pregnancy test before study participation AND is willing to take an additional pregnancy test during the study as appropriate and necessary, and as determined by the Medical Director of the study.
* Child and parent willing to give permission for the study team to contact the child's primary care physician, mental health clinician and /or mental health prescriber to communicate any changes in child's symptom status or medications as a result of participation in this research.

Exclusion Criteria

:• A history of cardiovascular disease, previous history of ECG abnormalities, syncope, exercise-induced cardiovascular symptoms, or any other unstable medical illness/allergy (i.e., seizure disorder) that in the opinion of the site Medical Director precludes enrollment in the study. A clinically significant history of Raynaud's disease is exclusionary.

* Autistic disorder, persons with intellectual disability (IQ ≤ 70), clinically significant (in the judgment of the site Medical Director) substance abuse disorder (within the past 30 days), bipolar I disorder, schizophrenia or other psychotic disorder, or major depressive disorder with symptoms that are severe enough (e.g. suicidality) that in the opinion of the site Medical Director excludes study participation.
* Concomitant Medications: Use of other psychiatric medications including extended release guanfacine (study drug) besides a stable dose of stimulants or atomoxetine for ADHD for the study duration is exclusionary for this protocol. All other medications will undergo discontinuation.
* Patients who are unable to comply with the study protocol.
* Females of childbearing age that are sexually active and not receiving a medically acceptable form of birth control and/or active pregnancy.
* Already taking Guanfacine Extended Release

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2019-12-03 (Actual)

PRIMARY OUTCOMES:
Changes in the Structured Trauma-Related Experiences and Symptoms Screener (STRESS) | Completed as part of the initial evaluation (T0), after drug dose has been determined to be stable and fixed (T1), and after completing the Mindfulness Therapy. (T2) (approximately 20 weeks in total)
  a self-report and observer-report instrument for youths 7-18 years that inventories 25 adverse childhood experiences and potentially traumatic events and assesses symptoms of post-traumatic stress disorder using the revised criteria published in DSM 5. Total score and DSM 5 domains B-E are included (intrusive symptoms, avoidance, cognitive-mood symptoms, arousal-reactivity symptoms and symptoms of dissociation).
Changes in theRetrospective-Modified Overt Aggression Scale (R-MOAS) | Completed as part of the initial evaluation (T0), after drug dose has been determined to be stable and fixed (T1), and after completing the Mindfulness Therapy. (T2)(approximately 20 weeks in total)
  (R-MOAS) assesses the frequency and severity of 16 aggressive behaviors over the past week in four areas: verbal aggression, physical aggression towards others, aggression toward oneself, and destruction or hostile misuse of property. Numeric weighting amplifies the seriousness of more harmful behaviors in the total score. Reliability and validity data on the instrument are published. A total score ≥ 24 is required to identify clinically significant aggression.
Changes in ADHD RS-IV | Completed as part of the initial evaluation (T0), after drug dose has been determined to be stable and fixed (T1), and after completing the Mindfulness Therapy. (T2)(approximately 20 weeks in total)
  An 18-item caregiver-completed rating scale developed to measure the behaviors of youths with ADHD
Changes in the Emotion Reactivity Scale (ERS) | Completed as part of the initial evaluation (T0), after drug dose has been determined to be stable and fixed (T1), and after completing the Mindfulness Therapy. (T2). Also at each medication management appointment(approximately 20 weeks in total)
  A 21-item self-report measure of emotion sensitivity, intensity, and persistence. The scale assesses emotional reactivity.
Youth Self Report (CBCL) | Completed at initial visit only (week 1)
  Assesses self-report functioning and internalizing and externalizing symptoms. The YSR contains social competence items and 112 items assessing self-reported symptoms.
Kaufman Brief Intelligence Test-2 | Completed by the adolescent at the initial visit only (week 1)
  The KBIT is normed for ages 4-90 years and yields a verbal IQ, non-verbal IQ, and full-scale IQ.

SECONDARY OUTCOMES:
Guanfacine Extended Release and Mindfulness Skills Therapy reducing traumatic stress | 20 weeks
  1. To measure whether Guanfacine Extended Release (GXR) 1-7 mg/daily compared to placebo will help diminish traumatic stress-related symptoms of concentration difficulties, aggression and anger, irritability, anxiety, fear, and depression in 12-17 year old youths who have experienced lifetime traumatic stress as assessed by clinician-reports, and observer- and self-reports on psychometrically validated rating scales.
Tolerance of Guanfacine Extended Release in subjects between the ages of 12-17 years old. | 20 weeks
  2. To measure how well 12-17 year-old children tolerate Guanfacine Extended Release (GXR) 1-7 mg/daily compared to placebo. Tolerance assessed by review of adverse events.
Clinical Global Impressions Improvement Scale | Completed ater drug dose has been determined to be stable and fixed (T1) and after completing the Mindfulness Therapy (T2) and each medication management visit.(approximately 20 weeks in total)
  The CGI-Improvement scale assesses patient overall improvement of symptoms compared with symptoms at study baseline. It is rated on a 7-point scale with scores ranging between 1 ("very much improved), 2 ("improved"), 3 ("minimally improved"), 4 ("no change from baseline") to 7 ("very much worse").
Clinical Global Impressions Severity Scale | Completed as part of the initial evaluation (T0), after drug dose has been determined to be stable and fixed (T1), and after completing the Mindfulness Therapy. (T2). Also at each medication management appointment(approximately 20 weeks in total)
  The CGI-Severity scale assesses the overall severity of a patient's psychiatric condition on a 7-point scale with scores ranging from 1 ("not ill") to 7 ("extremely severe").
Client Credibility Questionnaire (CCQ) | the CCQ will be administered to all youth and parents at the end of session one following presentation of the treatment rationale(approximately 20 weeks in total)
  measures youth and parent expectancies of treatment
Group Engagement Scale (GES) | At each of the Mindfulness Skills Therapy sessions if the subject is in group therapy.(approximately 10 weeks)
  20-item scale, that assesses youth attitude/satisfaction toward their specific group. Each item is rated on a 9-point scale. Groups can prompt different attitudes among group members which can affect the effectiveness of the intervention. The GES yields high alphas (>0.9). (Those receiving individual Mindfulness will not receive this scale)
The Screen for Child Anxiety Related Emotional Disorders (SCARED) | Completed as part of the initial evaluation (T0), after drug dose has been determined to be stable and fixed (T1), and after completing the Mindfulness Therapy. (T2). Also at each medication management visit(approximately 20 weeks in total)
  a 41-item self or observer-completed screen for child and adolescent anxiety disorders. Sub-scores assess for the presence of panic disorder, generalized anxiety disorder, separation anxiety disorder, social anxiety disorder, and significant school avoidance. Total scores ≥ 25 may indicate the presence of an anxiety disorder.
Patient Health Questionnaire (PHQ-9) | Completed as part of the initial evaluation (T0), after drug dose has been determined to be stable and fixed (T1), and after completing the Mindfulness Therapy. (T2) Also at each medication management visit(approximately 20 weeks in total)
  a 9-item self-report instrument assessing symptoms of depression. In clinically referred populations a total score ≥ 10 may identify clinically significant depression given the higher base-rate of depression in clinical populations than in epidemiological samples.

CONTACTS AND LOCATIONS:
Overall Officials: Asima F Zehgeer, MD, Principal Investigator — UConn Health
Locations (1):
- UConn Health, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
This is a multi center study being conducted in collaboration with Yale University. All shared data will be coded, with the code being held exclusively by the original contributing institute.